CLINICAL TRIAL: NCT05586789
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Phase III Clinical Trial to Examine the Clinical Efficacy and Safety of Ranquilon, 1 mg Tablets in Patients With Anxiety in Neurasthenia and Adjustment Disorders
Brief Title: A Study of the Efficacy and Safety of Ranquilon Tablets in Patients With Anxiety in Neurasthenia and Adjustment Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAN-03-03-2022
Record Dates: First submitted 2022-10-14; First posted 2022-10-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Anxiety; Neurasthenia; Adjustment Disorders
MeSH Terms: conditions — Anxiety Disorders; Neurasthenia; Adjustment Disorders | interventions — GB-115

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranquilon (Experimental): Study drug Ranquilon, tablets, 1 mg, 2 tablets 3 times a day (daily dose - 6 mg/day), daily, for 28 days
  Interventions: Drug: Ranquilon
- Placebo (Placebo Comparator): Placebo, tablets, 2 tablets 3 times a day, daily, for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranquilon — Two 1 mg tablets 3 times per day for 28 days
  Other Names: GB-115; 6-phenylhexanoyl)glycyl-L-tryptophan amide
  Arms: Ranquilon
Drug: Placebo — Two tablets 3 times per day for 28 days
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of Ranquilon, 1 mg tablets, at a dose of 6 mg/day compared to placebo for the treatment of patients with anxiety in neurasthenia and adjustment disorder.

An additional study objective was to evaluate the safety of Ranquilon, 1 mg tablets, at a dose of 6 mg/day compared to placebo in patients with anxiety in neurasthenia and adjustment disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 70
2. Presence of written consent to participate in the study in accordance with applicable law
3. Patients with anxiety and diagnoses based on ICD-10 criteria: neurasthenia (F48.0) or adjustment disorder (F43.2)
4. HARS anxiety scores of 18-24
5. Severity of asthenia on the Asthenia Self Assessment Scale (MFI-20) of more than 50 points
6. Hamilton Depression Assessment Scale (HAMD-17) score < 6
7. CGI-s scale score of at least 4
8. Negative pregnancy test for women of preserved reproductive potential
9. Consent to use effective contraception for the duration of the study and 30 days after completion (for women of unresolved reproductive potential and men)
10. Ability to understand the requirements for study participants, to give written consent to participate in the study (including the use and communication of patient health information relevant to the study) and to comply with the procedures of the study protocol

Exclusion Criteria:

1. Known intolerance to the active ingredient and/or excipients in the study drug/placebo of the study drug
2. Known presence of lactase deficiency, lactose intolerance, glucose-galactose malabsorption or galactose intolerance
3. Patients who require concomitant therapy prohibited in this study (MAO inhibitors, antidepressants, neuroleptics, anxiolytics and sedatives (including herbal), sleeping pills when used on a continuous basis), or have taken these drugs within the last month
4. Established or suspected alcohol/drug use at the time of screening or randomization, and/or a history of alcohol, drug or drug dependence
5. Presence of cancer, including a history of cancer (with the exception of a cured tumor with sustained remission for more than 5 years)
6. Presence of tuberculosis, including a history of tuberculosis
7. The presence of HIV, chronic viral hepatitis B/C, syphilis (including a history), or a positive test for HIV, hepatitis B/C, syphilis at screening
8. Patients with a diagnosis established on the basis of ICD-10 criteria: other anxiety disorders (F41)
9. Schizophrenia, schizoaffective, affective and panic disorders
10. Acute psychosis (endogenous-procedural, organic or somatogenic), including history
11. Organic lesions of the central nervous system of traumatic and alcoholic genesis
12. Postencephalitic syndrome
13. Brain tumors, including in the anamnesis
14. Degenerative diseases of the central nervous system (CNS), in particular, multiple sclerosis
15. Depression, including a history of depression
16. Generalized anxiety disorder, including a history
17. Suicidal thoughts or ideas; a history of suicide attempts
18. Epilepsy, seizures, including a history of seizures
19. Diabetes mellitus at the stage of decompensation
20. Established diagnosis of chronic kidney disease stage 3A or higher, or glomerular filtration rate (GFR) calculated by the Cockcroft-Gault formula = 59 ml/min/1.73 m2 or less
21. Established diagnosis of hepatic failure of any severity, or elevated ALT, AST or total bilirubin, urea >3 times the upper limit of normal values
22. Conditions after major surgical interventions, if less than six months have elapsed since the intervention
23. Chronic heart failure New York Heart Association (NYHA) functional class III-IV
24. Severe, decompensated, or unstable disease (any disease or condition that threatens the patient's life or worsens the patient's prognosis, or makes it impossible to perform a clinical trial in the patient)
25. Pregnant women, women breastfeeding, or women planning to become pregnant during the study and 30 days after study participation ends
26. Refusal by the patient to use approved contraception or to completely abstain from sexual intercourse during the entire period of study participation, beginning at Visit 0, and for 30 days after completion of study participation
27. Patient's current or planned participation in psychological or psychotherapeutic interventions designed to treat an anxiety disorder during the course of the clinical trial
28. Participation in any other clinical trial within 90 days prior to the screening period
29. Lack of willingness to cooperate on the part of the patient
30. Other reasons that, in the opinion of the investigator, prevent the patient from participating in the study or pose an unreasonable risk to the patient

Withdrawal Criteria:

1. Patient's desire to stop participating in the study (withdrawal of informed consent) Each patient has the right to stop participating in the study at any time without giving a reason. Withdrawal from the study will not affect the medical care provided to the patient in the future.
2. A decision by the research physician that the patient should be excluded is in the patient's own best interest
3. Patient refuses to cooperate with the investigator or is undisciplined
4. Causes/occurrence of situations during the study that threaten patient safety (e.g., hypersensitivity reactions, SAE, etc.)
5. Inclusion of a patient in the study with inclusion/inclusion criteria not met (prior to randomization)
6. Significant violation of the treatment regimen A significant violation is defined as a) skipping study drug/placebo for 2 consecutive full days or more, or b) taking, in total, < 80% or >120% of the full course (full course = 168 pills)
7. Positive pregnancy test
8. Confirmed diagnosis of COVID-19
9. Occurrence in the course of the study of other reasons that prevent the study according to the protocol
10. Death of a patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Change in patient status on the Hamilton Anxiety Rating Scale (HARS): Percentage of patients with a significant, i.e., 50% or greater reduction from baseline, in HARS anxiety levels on Day 29 ± 1 | Day 29 ± 1 of the study
  HARS scale includes 14 items, each of which is rated on the Likken scale. Of these, 13 items relate to the manifestation of anxiety in daily life, 14 items relate to the manifestation of anxiety during examinations. The sum of the scores may range from 0 to 56, with scores 0 to 7 corresponding to the absence of anxiety, 8 to 17 to the presence of symptoms of anxiety disorder, 18 to 24 to moderate severity of anxiety disorder, and 25 to 56 to severe severity of anxiety disorder.

SECONDARY OUTCOMES:
Proportion of patients with a significant, i.e., 50% or greater reduction in HARS anxiety level on Day 15 ± 1 (Visit 2) | Day 15 ± 1 of the study
  HARS scale includes 14 items, each of which is rated on the Likken scale. Of these, 13 items relate to the manifestation of anxiety in daily life, 14 items relate to the manifestation of anxiety during examinations. The sum of the scores may range from 0 to 56, with scores 0 to 7 corresponding to the absence of anxiety, 8 to 17 to the presence of symptoms of anxiety disorder, 18 to 24 to moderate severity of anxiety disorder, and 25 to 56 to severe severity of anxiety disorder.
Change in HARS anxiety level on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) compared to baseline | Day 15 ± 1 and Day 29 ± 1 of the study
  HARS scale includes 14 items, each of which is rated on the Likken scale. Of these, 13 items relate to the manifestation of anxiety in daily life, 14 items relate to the manifestation of anxiety during examinations. The sum of the scores may range from 0 to 56, with scores 0 to 7 corresponding to the absence of anxiety, 8 to 17 to the presence of symptoms of anxiety disorder, 18 to 24 to moderate severity of anxiety disorder, and 25 to 56 to severe severity of anxiety disorder.
Proportion of patients with HARS anxiety scores reduced to 17 or less on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) | Day 15 ± 1 and Day 29 ± 1 of the study
  HARS scale includes 14 items, each of which is rated on the Likken scale. Of these, 13 items relate to the manifestation of anxiety in daily life, 14 items relate to the manifestation of anxiety during examinations. The sum of the scores may range from 0 to 56, with scores 0 to 7 corresponding to the absence of anxiety, 8 to 17 to the presence of symptoms of anxiety disorder, 18 to 24 to moderate severity of anxiety disorder, and 25 to 56 to severe severity of anxiety disorder.
Time to decrease the HARS anxiety level to a score of 17 or less | Screening, Day 15 ± 1, Day 29 ± 1 of the study, the end of the study (Day 44 ± 1) or an early termination visit, whichever came first
  HARS scale includes 14 items, each of which is rated on the Likken scale. Of these, 13 items relate to the manifestation of anxiety in daily life, 14 items relate to the manifestation of anxiety during examinations. The sum of the scores may range from 0 to 56, with scores 0 to 7 corresponding to the absence of anxiety, 8 to 17 to the presence of symptoms of anxiety disorder, 18 to 24 to moderate severity of anxiety disorder, and 25 to 56 to severe severity of anxiety disorder.
Proportion of patients with significant and marked improvement as assessed by the physician (Clinical Global Impression - improvement (CGI-i) score 1 or 2) at Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) | Day 15 ± 1 and Day 29 ± 1 of the study
  The Clinical Global Impression Scale (CGI) includes two subscales: one for severity of symptoms and one for progression of symptoms with treatment. The first subscale is called Clinical Global Impression - severity (CGI-s) and the second subscale is Clinical Global Impression - improvement (CGI-i). CGI-s includes scores from 0 (healthy) to 7 (very severe); CGI-i includes scores from 1 (marked improvement) to 7 (marked deterioration)
Proportion of patients with a CGI-s score of 1 or 2 as assessed by the physician (healthy or borderline disorder) on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) | Day 15 ± 1 and Day 29 ± 1 of the study
  The Clinical Global Impression Scale (CGI) includes two subscales: one for severity of symptoms and one for progression of symptoms with treatment. The first subscale is called Clinical Global Impression - severity (CGI-s) and the second subscale is Clinical Global Impression - improvement (CGI-i). CGI-s includes scores from 0 (healthy) to 7 (very severe); CGI-i includes scores from 1 (marked improvement) to 7 (marked deterioration)
Time to significant or marked improvement - achieving a score of 1 or 2 on the CGI-i scale | Screening, Day 15 ± 1, Day 29 ± 1 of the study, or an early termination visit, whichever came first
  The Clinical Global Impression Scale (CGI) includes two subscales: one for severity of symptoms and one for progression of symptoms with treatment. The first subscale is called Clinical Global Impression - severity (CGI-s) and the second subscale is Clinical Global Impression - improvement (CGI-i). CGI-s includes scores from 0 (healthy) to 7 (very severe); CGI-i includes scores from 1 (marked improvement) to 7 (marked deterioration)
Time to decrease in severity of condition to 2 points or to 1 point or CGI-s scale | Screening, Day 15 ± 1, Day 29 ± 1 of the study, the end of the study (Day 44 ± 1) or an early termination visit, whichever came first
  The Clinical Global Impression Scale (CGI) includes two subscales: one for severity of symptoms and one for progression of symptoms with treatment. The first subscale is called Clinical Global Impression - severity (CGI-s) and the second subscale is Clinical Global Impression - improvement (CGI-i). CGI-s includes scores from 0 (healthy) to 7 (very severe); CGI-i includes scores from 1 (marked improvement) to 7 (marked deterioration)
Absolute value of the patient's CGI-i score by Days 15 ± 1 (Visit 2) and 29 ± 1 (Visit 3) | Day 15 ± 1 and Day 29 ± 1 of the study
  The Clinical Global Impression Scale (CGI) includes two subscales: one for severity of symptoms and one for progression of symptoms with treatment. The first subscale is called Clinical Global Impression - severity (CGI-s) and the second subscale is Clinical Global Impression - improvement (CGI-i). CGI-s includes scores from 0 (healthy) to 7 (very severe); CGI-i includes scores from 1 (marked improvement) to 7 (marked deterioration)
Change in patient severity on the CGI-s scale by Days 15 ± 1 (Visit 2) and 29 ± 1 (Visit 3) compared to baseline | Day 15 ± 1 and Day 29 ± 1 of the study
  The Clinical Global Impression Scale (CGI) includes two subscales: one for severity of symptoms and one for progression of symptoms with treatment. The first subscale is called Clinical Global Impression - severity (CGI-s) and the second subscale is Clinical Global Impression - improvement (CGI-i). CGI-s includes scores from 0 (healthy) to 7 (very severe); CGI-i includes scores from 1 (marked improvement) to 7 (marked deterioration)
Change in the Multidimensional Fatigue Fatigue Inventory (MFI-20) total score on Day 15 ± 1 (Visit 2) and 29 ± 1 (Visit 3) compared to baseline | Day 15 ± 1 and Day 29 ± 1 of the study
  The Multidimensional Fatigue Fatigue Inventory (MFI-20) provides a subjective quantitative assessment of the overall severity of asthenia and its various aspects. This scale consists of 20 items reflecting the main components of asthenic syndrome, such as: general asthenia, physical asthenia, mental asthenia, decreased activity and decreased motivation. The patient was given an opportunity to rate the mentioned items to his/her condition on a five-point scale. The score of the scale is the sum of the points of its individual constituent items and can vary in the range from 5 to 25 points. Normally, the total number of points should not exceed 30. If the total score on one of the subscales was higher than 12, this could be a preliminary ground for classifying the condition as an asthenic syndrome
Time to decrease the MFI-20 cumulative score to 30 points or less | Screening, Day 15 ± 1, Day 29 ± 1 of the study, or an early termination visit, whichever came first
  The Multidimensional Fatigue Fatigue Inventory (MFI-20) provides a subjective quantitative assessment of the overall severity of asthenia and its various aspects. This scale consists of 20 items reflecting the main components of asthenic syndrome, such as: general asthenia, physical asthenia, mental asthenia, decreased activity and decreased motivation. The patient was given an opportunity to rate the mentioned items to his/her condition on a five-point scale. The score of the scale is the sum of the points of its individual constituent items and can vary in the range from 5 to 25 points. Normally, the total number of points should not exceed 30. If the total score on one of the subscales was higher than 12, this could be a preliminary ground for classifying the condition as an asthenic syndrome
Time to decrease the MFI-20 cumulative score by 25% and 50% from baseline | Screening, Day 15 ± 1, Day 29 ± 1 of the study, or an early termination visit, whichever came first
  The Multidimensional Fatigue Fatigue Inventory (MFI-20) provides a subjective quantitative assessment of the overall severity of asthenia and its various aspects. This scale consists of 20 items reflecting the main components of asthenic syndrome, such as: general asthenia, physical asthenia, mental asthenia, decreased activity and decreased motivation. The patient was given an opportunity to rate the mentioned items to his/her condition on a five-point scale. The score of the scale is the sum of the points of its individual constituent items and can vary in the range from 5 to 25 points. Normally, the total number of points should not exceed 30. If the total score on one of the subscales was higher than 12, this could be a preliminary ground for classifying the condition as an asthenic syndrome
Proportion of patients with a 25% reduction in MFI-20 total score on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) from baseline | Day 15 ± 1 and Day 29 ± 1
  The Multidimensional Fatigue Fatigue Inventory (MFI-20) provides a subjective quantitative assessment of the overall severity of asthenia and its various aspects. This scale consists of 20 items reflecting the main components of asthenic syndrome, such as: general asthenia, physical asthenia, mental asthenia, decreased activity and decreased motivation. The patient was given an opportunity to rate the mentioned items to his/her condition on a five-point scale. The score of the scale is the sum of the points of its individual constituent items and can vary in the range from 5 to 25 points. Normally, the total number of points should not exceed 30. If the total score on one of the subscales was higher than 12, this could be a preliminary ground for classifying the condition as an asthenic syndrome
Proportion of patients with a 50% reduction in MFI-20 total score on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) from baseline | Day 15 ± 1 and Day 29 ± 1
  The Multidimensional Fatigue Fatigue Inventory (MFI-20) provides a subjective quantitative assessment of the overall severity of asthenia and its various aspects. This scale consists of 20 items reflecting the main components of asthenic syndrome, such as: general asthenia, physical asthenia, mental asthenia, decreased activity and decreased motivation. The patient was given an opportunity to rate the mentioned items to his/her condition on a five-point scale. The score of the scale is the sum of the points of its individual constituent items and can vary in the range from 5 to 25 points. Normally, the total number of points should not exceed 30. If the total score on one of the subscales was higher than 12, this could be a preliminary ground for classifying the condition as an asthenic syndrome
Proportion of patients with a decrease in their MFI-20 cumulative score to 30 on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) | Day 15 ± 1 and Day 29 ± 1
  The Multidimensional Fatigue Fatigue Inventory (MFI-20) provides a subjective quantitative assessment of the overall severity of asthenia and its various aspects. This scale consists of 20 items reflecting the main components of asthenic syndrome, such as: general asthenia, physical asthenia, mental asthenia, decreased activity and decreased motivation. The patient was given an opportunity to rate the mentioned items to his/her condition on a five-point scale. The score of the scale is the sum of the points of its individual constituent items and can vary in the range from 5 to 25 points. Normally, the total number of points should not exceed 30. If the total score on one of the subscales was higher than 12, this could be a preliminary ground for classifying the condition as an asthenic syndrome
Change in Spielberger personality anxiety level on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) compared to baseline | Day 15 ± 1 and Day 29 ± 1
  The Spielberger Questionnaire includes a series of statements describing personal and situational anxiety, the answers to which are scored from 1 (least severe or prolonged) to 4 (most severe or prolonged). The patient reads the statements and independently chooses the most appropriate frequency for each statement. When analyzing the results of the self-assessment, you should keep in mind that the overall total for each of the subscales may range from 20 to 80 points. The higher the total score, the higher the level of anxiety (situational or personal).
Change in situational anxiety levels on the Spielberger questionnaire on Day 15 ± 1 (Visit 2) and Day 29 ± 1 (Visit 3) compared to baseline | Day 15 ± 1 and Day 29 ± 1
  The Spielberger Questionnaire includes a series of statements describing personal and situational anxiety, the answers to which are scored from 1 (least severe or prolonged) to 4 (most severe or prolonged). The patient reads the statements and independently chooses the most appropriate frequency for each statement. When analyzing the results of the self-assessment, you should keep in mind that the overall total for each of the subscales may range from 20 to 80 points. The higher the total score, the higher the level of anxiety (situational or personal).
Safety and Tolerability: adverse event (AE) rate | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 44 ± 1 for each participant
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: AEs associated with the study drug | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 44 ± 1 for each participant
  Number and frequency of AEs or SAEs associated with the study drug
Safety and Tolerability: treatment discontinuation | From the date of screening (and signing informed consent form) to the end of the study or to an early termination visit, whichever came first, assessed up to day 44 ± 1 for each participant
  Percentage of patients who discontinued treatment due to the occurrence of AEs/SAEs
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | Screening, day 1, day 15, day 29, and day 44 of the study or on the early termination visit, whichever came first, within 44 days of study participation
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | Screening, day 1, day 15, day 29, and day 44 of the study or on the early termination visit, whichever came first, within 44 days of study participation
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | Screening, day 1, day 15, day 29, and day 44 of the study or on the early termination visit, whichever came first, within 44 days of study participation
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | Screening, day 1, day 15, day 29, and day 44 of the study or on the early termination visit, whichever came first, within 44 days of study participation
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | Screening, day 1, day 15, day 29, and day 44 of the study or on the early termination visit, whichever came first, within 44 days of study participation
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | Screening, day 1, day 15, day 29, and day 44 of the study or on the early termination visit, whichever came first, within 44 days of study participation
  Physical examination will follow the general rules of internal medicine: general examination, examination of mucous membranes and skin, including palpation of lymph nodes, evaluation of the musculoskeletal system, palpation, percussion, and auscultation of the main organ systems (cardiovascular, respiratory, digestive, and urinary systems) will be performed sequentially
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | Screening, day 29, or on the early termination visit, whichever came first, within 44 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | Screening, day 29, or on the early termination visit, whichever came first, within 44 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | Screening, day 29, or on the early termination visit, whichever came first, within 44 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | Screening, day 29, or on the early termination visit, whichever came first, within 44 days of study participation
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)
Safety and Tolerability: complete blood count - hemoglobin | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - hematocrit | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Hematocrit, %
Safety and Tolerability: complete blood count - red blood cells | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - white blood cells | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - platelets | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: complete blood count - lymphocytes | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Eosinophils, %
Safety and Tolerability: complete blood count - monocytes | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Basophils, %
Safety and Tolerability: complete blood count - neutrophils | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Neutrophils, % (segmented and stab)
Safety and Tolerability: blood test results - total cholesterol | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Total cholesterol in blood serum, mmol/L
Safety and Tolerability: blood test results - total protein | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - glucose | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - creatinine | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - alanine transaminase (ALT) | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  AST in blood serum, U/L
Safety and Tolerability: blood test results - total bilirubin | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - direct bilirubin | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Direct bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - alkaline phosphatase (ALP) | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  ALP in blood serum, U/L
Safety and Tolerability: blood test results - urea | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Urea in blood serum, mmol/L
Safety and Tolerability: urinalysis - color | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Color of the urine (yellow, brown, etc.)
Safety and Tolerability: urinalysis - transparency | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Transparency of the urine (transparent/cloudy)
Safety and Tolerability: urinalysis - specific gravity | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Specific gravity of the urine
Safety and Tolerability: urinalysis - pH | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  pH of the urine
Safety and Tolerability: urinalysis - glucose | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis - protein | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis - ketones | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Ketones in the urine (mmol/L)
Safety and Tolerability: urinalysis - urobilinogen | Screening, Day 29 or the early termination visit, whichever came first, within 44 days of study participation
  Urobilinogen in the urine (umol/L)

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Engels Psychiatric Hospital State Health Care Institution of the Ministry of Health of the Saratov Region, Engel's
  - State Budgetary Health Institution of Nizhny Novgorod Oblast "Clinical Psychiatric Hospital No. 1 of Nizhny Novgorod. Nizhny Novgorod", Nizhny Novgorod
  - Professors' Clinic LLC., Perm
  - Limited Liability Company "Research Center Eco-Security", Saint Petersburg
  - EosMED JSC, Saint Petersburg
  - Limited Liability Company "Energy of Health", Saint Petersburg
  - LLC "Aurora MedFort", Saint Petersburg
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg
  - Limited Liability Company "Meili", Saint Petersburg
  - Saratov City Psychoneurological Dispensary, Saratov

IPD SHARING:
Plan to Share IPD: Undecided